CLINICAL TRIAL: NCT02067481
Title: Effect of a Diet and Physical Activity Intervention on Body Weight and Nutritional Patterns in Overweight and Obese Breast Cancer Survivors
Brief Title: Effect of a Diet and Physical Activity Intervention in Breast Cancer Survivors
Acronym: PREDICOP-F
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREDICOP-F
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Survivors; Weight loss; Diet; Physical activity
MeSH Terms: conditions — Breast Neoplasms; Weight Loss; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm weight loss intervention (Experimental): This single-arm pre-post study, that involved one-hourly weekly diet sessions delivered by a dietician and 75-minute bi-weekly Physical Activity (AP) sessions of moderate-to-high intensity led by PA monitors, was offered to overweight and obese BC survivors shortly after treatment.
  Interventions: Behavioral: Weight loss intervention

INTERVENTIONS:
Behavioral: Weight loss intervention — This single-arm pre-post study, that involved one-hourly weekly diet sessions delivered by a dietician and 75-minute bi-weekly Physical Activity (PA) sessions of moderate-to-high intensity led by PA monitors, was offered to overweight and obese BC survivors shortly after treatment. Before and after the intervention, anthropometry, dietary information, Quality of Life (QoL) and cardiorespiratory fitness (CRF) were collected.
  Other Names: Dietary and Physical Activity Intervention

SUMMARY:
This is a single-arm pre-post pilot study, to assess changes in weight, quality of life and cardiorespiratory fitness after a diet and physical activity intervention in breast cancer survivors and to asses possible relation between these changes.

DETAILED DESCRIPTION:
Aim:

The present study assessed changes in weight, quality of life (QoL) and cardiorespiratory fitness (CRF) during a diet and physical activity (PA) intervention in breast cancer (BC) survivors and investigated the possible relation between these changes.

Methods:

The intervention of this 12-week single-arm pre-post pilot study involved group-based sessions: one-hour weekly diet sessions delivered by a dietician and 75-minute bi-weekly PA sessions of moderate-to-high intensity led by PA monitors. This intervention, designed to promote weight loss, targeted overweight/obese women who had completed treatment less than six months before recruitment. CRF and QoL were assessed before and after the intervention and compared using paired t-tests. Linear regression models, including CRF variables, weight change and participants' characteristics, were used to assess the independent association between change in CRF and change in QoL.

ELIGIBILITY:
Inclusion Criteria:

* Female patients from the Catalan Institute of Oncology
* Aged 18 to 75
* Body mass index (BMI) of 25 kg•m-2 or more
* Completed chemotherapy and/or radiotherapy for breast cancer during the 6 months preceding recruitment

Exclusion Criteria:

* First cancer, tumours of stage IIIB and above
* Morbid obesity (BMI ≥40 kg•m-2)
* Any condition that could not permit to follow the diet and PA intervention offered

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months
  Loss 3% of the initial weight

SECONDARY OUTCOMES:
Quality of life | 3 months
  EORTC QLQ-C30 and BR23 mean scores

OTHER OUTCOMES:
Biomarkers | 3 months
  Blood analysis: Biomarkers related to glucose, lipid profile, IGF1, reproductive hormones, leptin, adiponectin, carotenoids, inflammation markers, oxidative stress markers and hematologic parameters, will be analysed
Cardiorespiratory fitness | 3 months
  To determine peak oxygen uptake (VO2peak), an incremental cycle-ergometer test with monitoring ECG will be performed by exercise physiologists after a 24h period without physical activity in the Physiology Department of the University of Barcelona
Dietary habits | 3 months
  A validated food frequency questionnaire will be used, designed to capture dietary habits, 24-hour dietary recalls (covering week days and weekends) will be taken to calculate the patients' energy intake and nutritional profile.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Agudo, MsC PhD, Principal Investigator — Institut Catalá de Oncología
Locations (1):
- Instituto Catalá de Oncología, Barcelona, L´Hospitalet de Llobregat, Spain